CLINICAL TRIAL: NCT02208843
Title: An Open Label, Single-arm Phase IV Study to Assess the Efficacy and Safety of Afatinib as Second-line Therapy for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harbouring an EGFR Mutation (Del19 or L858R) Who Have Failed First-line Treatment With Platinum-based Chemotherapy
Brief Title: Afatinib as Second-line Therapy for Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.217; 2014-001077-14 (EudraCT Number)
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental): Afatinib tablet once daily until progression
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib tablet once daily until progression

SUMMARY:
The objectives of this single-arm, open-label trial are to assess the efficacy and safety of afatinib as second line treatment for patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harbouring a common EGFR mutation who have failed first-line platinum-based chemotherapy and to demonstrate that the efficacy and safety are comparable to the results seen in previous trials.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically confirmed diagnosis of Stage IIIB (with cytologically proven pleural effusion or pericardial effusion) or Stage IV adenocarcinoma of the lung. Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
2. Documented EGFR mutation (L858R and/or Deletion 19) with no other known EGFR mutation.
3. Measureable disease according to RECIST 1.1.
4. Radiologically confirmed progression or recurrence of disease during or following first line therapy with a platinum-based chemotherapy regimen.
5. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
6. Adequate organ function.

Exclusion criteria:

1. More than one line of prior therapy for disease.
2. Previously received less than 3 cycles of platinum-based chemotherapy due to toxicity and/or intolerance of treatment.
3. Previous treatment with any EGFR targeting Tyrosine Kinase Inhibitor (TKI) or antibody.
4. Known pre-existing interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (21):
- Egypt (3):
  - Clinical Research Center, Alexandria University Hospital, Alexandria
  - National Cancer Institute, Cairo University, Cairo
  - Kasr Al Ainy Hospital, Cairo
- Nilai Medical Centre, Kampung Baharu Nilai, Malaysia
- Philippines (2):
  - Baguio General Hospital and Medical Center, Baguio City
  - St. Luke's Medical Center, City of Taguig
- Poland (3):
  - University Clinical Center, Gdansk, Gdansk
  - Specialist Hospital, Szczecin-Zdunowo, Szczecin-Zdunowo
  - Oncol Centre M Sklodowska-Curie, Dept of Lung & Chest Cancer, Warsaw
- Romania (4):
  - Braila County Emergency Hospital, Medical Oncology, Brăila
  - Institute of Oncology 'Prof. Dr. Alexandru Trestioreanu', Bucharest
  - Sf. Nectarie Oncology Center, Craiova, Craiova
  - Regional Oncology Institute of Iasi, Medical Oncology, Iași
- Serbia (4):
  - Institute for Oncol & Radiol of Serbia, Clinic f. Med. Onco., Belgrade
  - Clinical Center of Serbia, Belgrade
  - Inst. for Pulm. Diseases of Vojvodine, Clinic f. Pulm. Oncol, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- Thailand (4):
  - Wattanosoth Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Songklanagarind Hospital, Songkhla

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, single-arm phase IV study to assess the efficacy and safety of Afatinib as second-line therapy for patients with locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) harbouring an Epidermal Growth Factor Receptor(EGFR) mutation (Del19 or L858R) who have failed first-line treatment with platinum-based chemotherapy.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Afatinib 40 mg: All patients received continuous daily treatment with Afatinib at a starting dose of 40 milligram (mg), treatment interruption and reduction scheme to 30 mg and then to 20 mg were permitted to manage treatment-related adverse events (AEs). Patients were orally administered with the film coated tablet once a day without food.
Period: Overall Study
Arm/Group | Afatinib 40 mg
Started (Patients entered the study and all received at least 1 dose of afatinib) | 60
Completed | 0
Not Completed | 60
Not completed — Clinical symptoms of progression | 2
Not completed — Progression disease according to RECIST | 24
Not completed — Adverse Event | 12
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Switched to commercial afatinib | 20

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
  Years | 59.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of subjects is categorized as Male or Female. Population: Treated Set (TS): The TS included all patients who were documented to have taken at least 1 dose of afatinib.
  Participants
    Female | 33
    Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of subjects is categorized for race data. Ethnicity data were not collected for this study. Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
  Participants
    American Indian or Alaska Native | 0
    Asian | 19
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 41
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumour Response (Complete Response [CR], Partial Response [PR]) as Assessed by the Investigator According to the RECIST Version 1.1
Description: As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by Magnetic resonance imaging (MRI): Complete Response (CR), disappearance of all target lesions; Partial Response (PR), =30% decrease in the sum of the longest diameter of target lesions
Time Frame: Post baseline tumour-imaging was performed at every 8 weeks until Week 56 and then every 12 weeks; up to 802 days
Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 60
Percentage of participants | 50 [36.8 to 63.2]

2. Secondary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator According to RECIST 1.1.
Description: Progression-free survival (PFS) is the time from treatment start to disease progression (or death if the patient died before progression). PFS as assessed based on investigator review according to the response evaluation criteria in solid tumours (RECIST) version 1.1.
Time Frame: Post baseline tumour-imaging was performed at every 8 weeks until Week 56 and then every 12 weeks; up to 802 days
Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 60
Months | 10.94 [6.44 to 13.20]

3. Secondary Outcome: Disease Control (CR, PR, Stable Disease [SD]) as Assessed by the Investigator According to RECIST 1.1
Description: As Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), =30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
Time Frame: Post baseline tumour-imaging was performed at every 8 weeks until Week 56 and then every 12 weeks; up to 802 days
Population: Treated Set (TS): The TS includes all patients who were documented to have taken at least 1 dose of afatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 60
Percentage of participants | 83.3 [71.5 to 91.7]

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 830 days
Arm/Group | Afatinib 40 mg
All-Cause Mortality (participants affected / at risk) | 11/60
Serious Adverse Events (participants affected / at risk) | 21/60
Other Adverse Events (participants affected / at risk) | 56/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=60)
Cardiac arrest (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Pneumonia (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=60)
Anaemia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 44
Nausea (Gastrointestinal disorders) | 12
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 6
Paronychia (Infections and infestations) | 14
Gamma-glutamyltransferase increased (Investigations) | 5
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 5
Nail pitting (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 18
Fatigue (General disorders) | 9
Mucosal inflammation (General disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT02208843/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT02208843/SAP_001.pdf